CLINICAL TRIAL: NCT05756985
Title: Improving Understanding of Glioblastoma Through Preservation of Biologically Active Brain Tissue (PRESERVE GBM)
Brief Title: Improving Understanding of Glioblastoma Through Preservation of Biologically Active Brain Tissue
Status: Recruiting | Type: Observational
Sponsor: Baptist Health South Florida (Other)
Collaborators: Miami Cancer Institute (Other); Nico Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022-SPEC-AHL-001
Record Dates: First submitted 2023-02-24; First posted 2023-03-07 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Glioblastoma; Glioblastoma Multiforme; Gliosarcoma
Keywords: specimen banking
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood: 50 mL (less than 4 tablespoons) Glioblastoma tissue: three geographically distinct samples from the same tumor, about 10 cubic centimeters in volume
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Glioblastoma: Surgical tumor resection as standard of care and specimen collection
  Interventions: Procedure: Specimen Collection

INTERVENTIONS:
Procedure: Specimen Collection — Collect and preserve glioblastoma tissue for exploratory analyses to generate hypotheses for future studies.

SUMMARY:
To collect and preserve glioblastoma tissue during standard of care tumor resection surgery and blood for future molecular and genetic testing. Tissue for research will be collected from three different regions within the same tumor to study how these regions differ in their structure, DNA, and RNA and also to compare the data obtained from this testing to imaging data found in the medical record. The goal of this study is to help us better understand what the glioblastoma tumor tissue looks like and how it functions. This understanding can lead to new therapies for the treatment of glioblastoma in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Have the appearance of high-grade glioma on magnetic resonance (MR) imaging if allowed to consent and will undergo the procedure if the frozen is consistent with glioblastoma or gliosarcoma OR Patients with a history of histologically confirmed diagnosis of World Health Organization Grade glioblastoma or gliosarcoma that are undergoing repeat resection of a recurrent tumor as identified on preoperative MR imaging
2. Aged ≥ 18 years old
3. Contrast-enhancing tumor volume of at least 10 cc on the preoperative, volumetric MRI within 1 month prior to surgery
4. Provision of signed and dated informed consent form by participant or legally authorized representative (LAR), if applicable

Exclusion Criteria:

1. Has a history or current evidence of any medical condition, therapy, or laboratory abnormality that might confound the results of the study or is not in the best interest of the participant, in the opinion of the treating investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with GBM or gliosarcoma undergoing standard of care tumor resection surgery.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Number of glioblastoma (GBM) samples for analysis | 2 years
  Total number of GBM samples collected and preserved for analysis

CONTACTS AND LOCATIONS:
Overall Officials: Manmeet S Ahluwalia, M.D., Principal Investigator — Miami Cancer Institute at Baptist Health, Inc.
Locations (1):
- Miami Cancer Institute at Baptist Health, Inc., Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] GLASS Consortium. Glioma through the looking GLASS: molecular evolution of diffuse gliomas and the Glioma Longitudinal Analysis Consortium. Neuro Oncol. 2018 Jun 18;20(7):873-884. doi: 10.1093/neuonc/noy020. PMID 29432615
- [Background] Kumar A, Boyle EA, Tokita M, Mikheev AM, Sanger MC, Girard E, Silber JR, Gonzalez-Cuyar LF, Hiatt JB, Adey A, Lee C, Kitzman JO, Born DE, Silbergeld DL, Olson JM, Rostomily RC, Shendure J. Deep sequencing of multiple regions of glial tumors reveals spatial heterogeneity for mutations in clinically relevant genes. Genome Biol. 2014 Dec 3;15(12):530. doi: 10.1186/s13059-014-0530-z. PMID 25608559
- [Background] Lee JK, Wang J, Sa JK, Ladewig E, Lee HO, Lee IH, Kang HJ, Rosenbloom DS, Camara PG, Liu Z, van Nieuwenhuizen P, Jung SW, Choi SW, Kim J, Chen A, Kim KT, Shin S, Seo YJ, Oh JM, Shin YJ, Park CK, Kong DS, Seol HJ, Blumberg A, Lee JI, Iavarone A, Park WY, Rabadan R, Nam DH. Spatiotemporal genomic architecture informs precision oncology in glioblastoma. Nat Genet. 2017 Apr;49(4):594-599. doi: 10.1038/ng.3806. Epub 2017 Mar 6. PMID 28263318
- [Background] Prasanna P, Patel J, Partovi S, Madabhushi A, Tiwari P. Radiomic features from the peritumoral brain parenchyma on treatment-naive multi-parametric MR imaging predict long versus short-term survival in glioblastoma multiforme: Preliminary findings. Eur Radiol. 2017 Oct;27(10):4188-4197. doi: 10.1007/s00330-016-4637-3. Epub 2016 Oct 24. PMID 27778090
- See also: Miami Cancer Institute — http://cancer.baptisthealth.net